CLINICAL TRIAL: NCT06346626
Title: To Evaluate the Consistency and Repeatability of Portable Automatic Optometry 2-WINS for Cycloplegic Optometry in Adolescents and Children
Status: Completed | Type: Observational
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2WIN-S2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-03

CONDITIONS: Optometry
Keywords: Cycloplegia; 2WIN-S; ARK-1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myopia, also known as short-sightedness or near-sightedness, is a prevalent condition that typically emerges during childhood and early adulthood. It occurs when the eye elongates excessively, causing images of distant objects to focus in front of the retina, leading to blurred distance vision. The number of people with myopia is increasing every year, reaching half of the world's population by 2050. The global potential productivity loss due to uncorrected refractive errors was $244 billion in 2015. Due to the strong association between high myopia and pathological changes in the choroid, retina, and sclera, leading to irreversible vision loss, and the fact that correcting the refractive error does not halt the progression of pathology, the prevention of myopia, especially high myopia, has emerged as a crucial international public health concern. In ocular examinations of children under noncycloplegic conditions, the influence of accommodation cannot be disregarded.

Cycloplegic refraction is widely regarded as the gold standard in epidemiological assessment of refractive errors in pediatric populations. Moreover, due to children's decreased cooperation and unreliable responses, subjective refraction tests are less valued, and objective tests under cycloplegia are preferred. The portable vision screener 2WIN-S is a binocular tool that detects various ocular abnormalities and measures the refraction of both eyes. Along with measuring phorias/tropias in prismatic diopters and objective refraction in the range of -15D to +15D, 2WIN-S also captures additional features.

This study employed the cycloplegic condition to measurements using 2WIN-S, ARK-1 and subjective testing, we wanted to test the reliability and accuracy of 2WIN-S.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 18 years old;
* The best corrected visual acuity is better than 0.1 (logmar);
* Patients undergoing eye mydriasis examination in the outpatient department of our hospital;
* Volunteer to participate in the study.

Exclusion Criteria:

* The subject who can not cooperate to complete the inspection;
* Have other eye diseases that cannot be dilated (such as angle-closure glaucoma, shallow front, etc.;
* Have other conditions that affect eye refraction, such as strabismus and previous eye surgery;
* Investigate other conditions that the doctor thinks should not be involved.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Refractive errors in children and adolescents
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The optometric result (2WIN-S) | One day
  The optometric result of 2WIN-S

SECONDARY OUTCOMES:
The optometric result(ARK-1) | One day
  The optometric result between 2WIN-S and ARK-1
The optometric result(subjective refraction) | One day
  The optometric result between 2WIN-S and subjective refraction

CONTACTS AND LOCATIONS:
Locations (1):
- He Eye Specialist Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
For reasonable requests, please contact the corresponding author to obtain data

REFERENCES:
- [Background] Baird PN, Saw SM, Lanca C, Guggenheim JA, Smith Iii EL, Zhou X, Matsui KO, Wu PC, Sankaridurg P, Chia A, Rosman M, Lamoureux EL, Man R, He M. Myopia. Nat Rev Dis Primers. 2020 Dec 17;6(1):99. doi: 10.1038/s41572-020-00231-4. PMID 33328468
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Naidoo KS, Fricke TR, Frick KD, Jong M, Naduvilath TJ, Resnikoff S, Sankaridurg P. Potential Lost Productivity Resulting from the Global Burden of Myopia: Systematic Review, Meta-analysis, and Modeling. Ophthalmology. 2019 Mar;126(3):338-346. doi: 10.1016/j.ophtha.2018.10.029. Epub 2018 Oct 17. PMID 30342076
- [Background] Magome K, Morishige N, Ueno A, Matsui TA, Uchio E. Prediction of cycloplegic refraction for noninvasive screening of children for refractive error. PLoS One. 2021 Mar 15;16(3):e0248494. doi: 10.1371/journal.pone.0248494. eCollection 2021. PMID 33720956
- [Background] Morgan IG, Iribarren R, Fotouhi A, Grzybowski A. Cycloplegic refraction is the gold standard for epidemiological studies. Acta Ophthalmol. 2015 Sep;93(6):581-5. doi: 10.1111/aos.12642. Epub 2015 Jan 18. PMID 25597549
- [Background] Paff T, Oudesluys-Murphy AM, Wolterbeek R, Swart-van den Berg M, de Nie JM, Tijssen E, Schalij-Delfos NE. Screening for refractive errors in children: the plusoptiX S08 and the Retinomax K-plus2 performed by a lay screener compared to cycloplegic retinoscopy. J AAPOS. 2010 Dec;14(6):478-83. doi: 10.1016/j.jaapos.2010.09.015. PMID 21168070
- [Background] Wilson LB, Melia M, Kraker RT, VanderVeen DK, Hutchinson AK, Pineles SL, Galvin JA, Lambert SR. Accuracy of Autorefraction in Children: A Report by the American Academy of Ophthalmology. Ophthalmology. 2020 Sep;127(9):1259-1267. doi: 10.1016/j.ophtha.2020.03.004. Epub 2020 Apr 18. PMID 32317177
- [Background] Hashemi H, Khabazkhoob M, Asharlous A, Soroush S, Yekta A, Dadbin N, Fotouhi A. Cycloplegic autorefraction versus subjective refraction: the Tehran Eye Study. Br J Ophthalmol. 2016 Aug;100(8):1122-7. doi: 10.1136/bjophthalmol-2015-307871. Epub 2015 Nov 5. PMID 26541436